CLINICAL TRIAL: NCT01326325
Title: Study of the Efficiency of the Ketamine With Low Analgesic Doses, in Association With High Opioids, in the Treatment of the Rebels Pains, in Palliative Phase of the Cancerous Disease
Brief Title: Efficacy of Low Analgesic Doses of Ketamine Associated With Opioids in Refractory Cancer Pain Treatment
Acronym: KEPAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P081242
Record Dates: First submitted 2011-03-22; First posted 2011-03-30 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Pain
Keywords: Cancer; Refractory pain; Uncontrolled pain; Ketamine
MeSH Terms: conditions — Pain; Neoplasms; Pain, Intractable | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (Experimental): Ketamine PANFARMA
  Interventions: Drug: Ketamine
- Not Ketamine (Placebo Comparator): NaCl
  Interventions: Drug: NaCl

INTERVENTIONS:
Drug: Ketamine — Drip continues of ketamine in intravenous injection included posology enters 0,5mg/kg /day and 2mg/kg/day during 4 days
  Arms: Ketamine
Drug: NaCl — Drip continues of NaCl 0,9% in intravenous injection during 4 days
  Arms: Not Ketamine

SUMMARY:
Long-term opioid therapy is commonly administered for the management of severe cancer pain. Increasing doses of opioids are titrated against effects until analgesia is achieved or intolerable adverse effects occur. Ketamine, an N-methyl-D-aspartate (NMDA) receptor antagonist, has been reported to improve analgesia in patients with uncontrolled pain receiving high doses of opioids. This study aims at determining the effectiveness of ketamine as an adjuvant to opioids in relieving cancer pain.

DETAILED DESCRIPTION:
Main objective:

To show that low analgesic doses of ketamine in intravenous infusion during 4 days associated with opioids better relieve refractory cancer pain than opioids without ketamine.

This study is a prospective study, multicenter (11 centres), consisting of 3 phases:

* a randomized controlled double blind phase of 5 days with 2 parallel groups of 38 patients each : ketamine (in association with high opioids), in intravenous injection during 4 days, versus placebo (in association with high opioids), in intravenous injection during 4 days ;
* an open-label phase of maximum 4 days, during which the ketamine Panpharma® is administered in intravenous infusion to the hospitalized patients who are still having uncontrolled pain persisting or recurrent ;
* an observational phase : starting at the discharge of the patient, of a maximal period of 6 months.The inclusion period is during 18 months, the total duration of the study is 2 years.

  76 patients are expected: 38 will be treated with opioids and ketamine; 38 will be treated with opioids and a placebo.

Success is defined by a decrease of the daily pain score of 50 % after 4 days. The expected rate of success in the placebo group is 10 % whereas the expected rate of success in the ketamine group is 30 %.

Primary outcome (pain score on a 11-point numerical scale) will be evaluated everyday as well as secondary outcomes (patient and clinician global impression of change, opioid consumption, adverse reactions, patient satisfaction on pain relief, sleep interference score).

Vital parameters (cardiac frequency, respiratory frequency and arterial blood pressure) will be checked everyday, many times a day : every hour for the four hours after the beginning of the treatment and then, every four hours ; every hour for the two hours following a dose shift).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized cancer patients (informed and conscious of the cancer diagnostic)
* Undergoing opioid treatment for 15 days at least
* Refractory pain (score higher than 5 on an 10-point numerical pain rating scale)
* Ability to score pain on a numerical pain rating scale
* Patient written agreement

Exclusion Criteria:

* Ketamine contraindications
* Methadone or other NMDA-antagonist treatment
* Karnofsky index under 10
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-07; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The percentage of reduction of the daily average score of painful intensity after 4 days of treatment (to J4), with regard to the basic value to J0 | 4 days
  The daily average score of painful intensity being the score of painful intensity of the previous 24 hours, determined by the patient on a digital scale(ladder) validated from 0 to 10

SECONDARY OUTCOMES:
Patient Global Impression of Change/ Clinical Global Impression of Change | 4 days
Daily sleep interference score | 4 days
Patient satisfaction of pain relief | 4 days
Opioids consumption | 4 days
Evaluate the adverse effects of opioids-ketamine association versus opioids-placebo | 4 days
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie ROSTAING-RIGATTIERI, MD, Principal Investigator — Center of Evaluation and Treatment of the pain - Saint-Antoine Hospital
Locations (1):
- Center of Evaluation and Treatment of the pain - Saint-Antoine Hospital, Paris, Île-de-France Region, France

REFERENCES:
- [Background] DOMINO EF, CHODOFF P, CORSSEN G. PHARMACOLOGIC EFFECTS OF CI-581, A NEW DISSOCIATIVE ANESTHETIC, IN MAN. Clin Pharmacol Ther. 1965 May-Jun;6:279-91. doi: 10.1002/cpt196563279. No abstract available. PMID 14296024
- [Background] Clements JA, Nimmo WS. Pharmacokinetics and analgesic effect of ketamine in man. Br J Anaesth. 1981 Jan;53(1):27-30. doi: 10.1093/bja/53.1.27. PMID 7459184
- [Background] Yamamura T, Harada K, Okamura A, Kemmotsu O. Is the site of action of ketamine anesthesia the N-methyl-D-aspartate receptor? Anesthesiology. 1990 Apr;72(4):704-10. doi: 10.1097/00000542-199004000-00021. PMID 1969718
- [Background] Franks NP, Lieb WR. Molecular and cellular mechanisms of general anaesthesia. Nature. 1994 Feb 17;367(6464):607-14. doi: 10.1038/367607a0. PMID 7509043
- [Background] Jacox A, Carr DB, Payne R. New clinical-practice guidelines for the management of pain in patients with cancer. N Engl J Med. 1994 Mar 3;330(9):651-5. doi: 10.1056/NEJM199403033300926. No abstract available. PMID 7508094
- [Background] Krakowski I, Theobald S, Balp L, Bonnefoi MP, Chvetzoff G, Collard O, Collin E, Couturier M, Delorme T, Duclos R, Eschalier A, Fergane B, Larue F, Magnet M, Minello C, Navez ML, Richard A, Richard B, Rostaing-Rigattieri S, Rousselot H, Santolaria N, Torloting G, Toussaint S, Vuillemin N, Wagner JP, Fabre N; FNCLCC. Summary version of the Standards, Options and Recommendations for the use of analgesia for the treatment of nociceptive pain in adults with cancer (update 2002). Br J Cancer. 2003 Aug;89 Suppl 1(Suppl 1):S67-72. doi: 10.1038/sj.bjc.6601086. No abstract available. PMID 12915905
- [Background] Rostaing-Rigattieri S, Rousselot H, Krakowski I, Theobald S, Collin E, Vuillemin N, Balp L, Torloting G, Fergane B, Richard B, Duclos R, Eschalier A, Delorme T, Minello C, Toussaint S, Richard A, Magnet M, Chvetzoff G, Larue F, Navez ML, Collard O, Bonnefoi MP, Couturier M, Santolaria N, Wagner JP, Fabre N. [Standards, options and recommendations for the use of medical analgesics for the treatment of pain arising from excess nociception in adults with cancer (update 2002): opioid analgesics with the exception of morphine by mouth and the rotation]. Bull Cancer. 2003 Aug-Sep;90(8-9):795-806. French. PMID 14609771
- [Background] Eide PK, Stubhaug A, Stenehjem AE. Central dysesthesia pain after traumatic spinal cord injury is dependent on N-methyl-D-aspartate receptor activation. Neurosurgery. 1995 Dec;37(6):1080-7. doi: 10.1227/00006123-199512000-00007. PMID 8584148
- [Background] Backonja M, Arndt G, Gombar KA, Check B, Zimmermann M. Response of chronic neuropathic pain syndromes to ketamine: a preliminary study. Pain. 1994 Jan;56(1):51-57. doi: 10.1016/0304-3959(94)90149-X. PMID 8159441
- [Background] Max MB, Byas-Smith MG, Gracely RH, Bennett GJ. Intravenous infusion of the NMDA antagonist, ketamine, in chronic posttraumatic pain with allodynia: a double-blind comparison to alfentanil and placebo. Clin Neuropharmacol. 1995 Aug;18(4):360-8. doi: 10.1097/00002826-199508000-00008. PMID 8665549
- [Background] Felsby S, Nielsen J, Arendt-Nielsen L, Jensen TS. NMDA receptor blockade in chronic neuropathic pain: a comparison of ketamine and magnesium chloride. Pain. 1996 Feb;64(2):283-291. doi: 10.1016/0304-3959(95)00113-1. PMID 8740606
- [Background] Nikolajsen L, Hansen CL, Nielsen J, Keller J, Arendt-Nielsen L, Jensen TS. The effect of ketamine on phantom pain: a central neuropathic disorder maintained by peripheral input. Pain. 1996 Sep;67(1):69-77. doi: 10.1016/0304-3959(96)03080-1. PMID 8895233
- [Background] Eide PK, Stubhaug A. Relief of glossopharyngeal neuralgia by ketamine-induced N-methyl-aspartate receptor blockade. Neurosurgery. 1997 Aug;41(2):505-8. doi: 10.1097/00006123-199708000-00043. PMID 9257324
- [Background] Kanamaru T, Saeki S, Katsumata N, Mizuno K, Ogawa S, Suzuki H. [Ketamine infusion for control of pain in patients with advanced cancer]. Masui. 1990 Oct;39(10):1368-71. Japanese. PMID 2255043
- [Background] Oshima E, Tei K, Kayazawa H, Urabe N. Continuous subcutaneous injection of ketamine for cancer pain. Can J Anaesth. 1990 Apr;37(3):385-6. doi: 10.1007/BF03005598. No abstract available. PMID 2322977
- [Background] Sosnowski M. Pain management: physiopathology, future research and endpoints. Support Care Cancer. 1993 Mar;1(2):79-88. doi: 10.1007/BF00366900. PMID 8143105
- [Background] Notcutt WG. Transporting patients with overwhelming pain. Anaesthesia. 1994 Feb;49(2):145-7. doi: 10.1111/j.1365-2044.1994.tb03373.x. PMID 8129125
- [Background] Clark JL, Kalan GE. Effective treatment of severe cancer pain of the head using low-dose ketamine in an opioid-tolerant patient. J Pain Symptom Manage. 1995 May;10(4):310-4. doi: 10.1016/0885-3924(95)00010-V. PMID 7541437
- [Background] Muller A, Lemos D. [Cancer pain: beneficial effect of ketamine addition to spinal administration of morphine-clonidine-lidocaine mixture]. Ann Fr Anesth Reanim. 1996;15(3):271-6. doi: 10.1016/s0750-7658(96)80005-0. French. PMID 8758581
- [Background] Yang CY, Wong CS, Chang JY, Ho ST. Intrathecal ketamine reduces morphine requirements in patients with terminal cancer pain. Can J Anaesth. 1996 Apr;43(4):379-83. doi: 10.1007/BF03011718. PMID 8697554
- [Background] Ashby MA, Martin P, Jackson KA. Opioid substitution to reduce adverse effects in cancer pain management. Med J Aust. 1999 Jan 18;170(2):68-71. doi: 10.5694/j.1326-5377.1999.tb126885.x. PMID 10026686
- [Background] Lauretti GR, Lima IC, Reis MP, Prado WA, Pereira NL. Oral ketamine and transdermal nitroglycerin as analgesic adjuvants to oral morphine therapy for cancer pain management. Anesthesiology. 1999 Jun;90(6):1528-33. doi: 10.1097/00000542-199906000-00005. PMID 10360847
- [Background] Fine PG. Low-dose ketamine in the management of opioid nonresponsive terminal cancer pain. J Pain Symptom Manage. 1999 Apr;17(4):296-300. doi: 10.1016/s0885-3924(98)00144-4. PMID 10203883
- [Background] Bell RF. Low-dose subcutaneous ketamine infusion and morphine tolerance. Pain. 1999 Oct;83(1):101-3. doi: 10.1016/s0304-3959(99)00096-2. PMID 10506678
- [Background] Lloyd-Williams M. Ketamine for cancer pain. J Pain Symptom Manage. 2000 Feb;19(2):79-80. doi: 10.1016/s0885-3924(99)00142-6. No abstract available. PMID 10766572
- [Background] Mercadante S, Arcuri E, Tirelli W, Casuccio A. Analgesic effect of intravenous ketamine in cancer patients on morphine therapy: a randomized, controlled, double-blind, crossover, double-dose study. J Pain Symptom Manage. 2000 Oct;20(4):246-52. doi: 10.1016/s0885-3924(00)00194-9. PMID 11027905
- [Background] Berger JM, Ryan A, Vadivelu N, Merriam P, Rever L, Harrison P. Ketamine-fentanyl-midazolam infusion for the control of symptoms in terminal life care. Am J Hosp Palliat Care. 2000 Mar-Apr;17(2):127-34. doi: 10.1177/104990910001700213. PMID 11406957
- [Background] Jackson K, Ashby M, Martin P, Pisasale M, Brumley D, Hayes B. "Burst" ketamine for refractory cancer pain: an open-label audit of 39 patients. J Pain Symptom Manage. 2001 Oct;22(4):834-42. doi: 10.1016/s0885-3924(01)00340-2. PMID 11576800
- [Background] McQueen AL, Baroletti SA. Adjuvant ketamine analgesia for the management of cancer pain. Ann Pharmacother. 2002 Oct;36(10):1614-9. doi: 10.1345/aph.1A256. PMID 12243612
- [Background] Kannan TR, Saxena A, Bhatnagar S, Barry A. Oral ketamine as an adjuvant to oral morphine for neuropathic pain in cancer patients. J Pain Symptom Manage. 2002 Jan;23(1):60-5. doi: 10.1016/s0885-3924(01)00373-6. PMID 11779670
- [Background] Persson J, Axelsson G, Hallin RG, Gustafsson LL. Beneficial effects of ketamine in a chronic pain state with allodynia, possibly due to central sensitization. Pain. 1995 Feb;60(2):217-222. doi: 10.1016/0304-3959(94)00139-6. PMID 7784107
- [Background] Cherry DA, Plummer JL, Gourlay GK, Coates KR, Odgers CL. Ketamine as an adjunct to morphine in the treatment of pain. Pain. 1995 Jul;62(1):119-121. doi: 10.1016/0304-3959(95)00010-P. PMID 7478701
- [Background] Shimoyama N, Shimoyama M, Inturrisi CE, Elliott KJ. Ketamine attenuates and reverses morphine tolerance in rodents. Anesthesiology. 1996 Dec;85(6):1357-66. doi: 10.1097/00000542-199612000-00017. PMID 8968183
- [Background] Bell R, Eccleston C, Kalso E. Ketamine as an adjuvant to opioids for cancer pain. Cochrane Database Syst Rev. 2003;(1):CD003351. doi: 10.1002/14651858.CD003351. PMID 12535471